CLINICAL TRIAL: NCT03548610
Title: Efficacy and Safety of a Nanofat-seeded Biological Scaffold in Healing Lower Limb Surgical Defects: A Randomized, Controlled Study
Brief Title: Efficacy and Safety of a Nanofat-seeded Biological Scaffold in Healing Lower Limb Surgical Defects
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: None of the screened subjects were interested / eligible for enrollment.
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Abigail Waldman,M.D., MOHS Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018P001086
Record Dates: First submitted 2018-05-17; First posted 2018-06-07 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Wound of Skin; Non-melanoma Skin Cancer; Skin Graft Complications; Wound of Lower Leg; Wound of Knee
Keywords: nanofat; tumor defect

STUDY DESIGN:
Intervention Model Description: Nanofat is obtained via lipoaspiration of 10cc of fat from abdomen under moderate local tumescent anesthesia w/ saline. Cannula access point is anesthetized by local lidocaine infiltration. Lipoaspirate is processed into the nanofat using the Tonnard method, after 3-minute decantation. Aspiration is performed using a multihole 3mm cannula. Wound margin + bed is treated w/ topical & local injections of nanofat, then covered w/ a biological scaffold, the inferior surface of which is soaked in nanofat; scaffold is fixed w/ external dressings or resorbable sutures; external covering includes polyurethane film & 3 layers of dressings. Topical application creates a fine <1mm nanofat layer. Scaffold (Puracol Plus) is left in place to integrate w/ surrounding skin, while external dressings changed at 7 & 15 days. Lipoaspirate donor site needs mild to moderate compression for 24 hours & suture removal (if not absorbed) at 7 days.
Who Masked: Outcomes Assessor
Masking Description: Blinded physician will evaluate standardized photographs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nanofat-seeded biological scaffold on surgical defect (Experimental): Nanofat is obtained via lipoaspiration of 10cc of fat from abdomen under moderate local tumescent anesthesia w/ saline. Cannula access point is anesthetized by local lidocaine infiltration. Lipoaspirate is processed into nanofat using the Tonnard method, after 3-minute decantation. Aspiration is performed using a multihole 3mm cannula. Wound margin + bed is treated w/ topical & local injections of nanofat, then covered w/ a biological scaffold, the inferior surface of which is soaked in nanofat; scaffold is fixed w/ external dressings or resorbable sutures; external covering includes polyurethane film & 3 layers of dressings. Topical application creates a fine <1mm nanofat layer. Scaffold (Puracol Plus) is left in place to integrate w/ surrounding skin, while external dressings changed at 7 & 15 days. Lipoaspirate donor site needs mild to moderate compression for 24 hours & suture removal (if not absorbed) at 7 days.
  Interventions: Other: Nanofat-seeded biological scaffold on surgical defect
- Standard of Care dressings (No Intervention): Immediately after surgical resection, each patient will be treated following the SOC, therefore with a local skin flap, rather than with a skin graft, based on surgeon assessment. Sutures, and moulage, if present, will be removed at 7 days and patient instructed to apply a daily silicone cream and sunscreen for 2 months.

INTERVENTIONS:
Other: Nanofat-seeded biological scaffold on surgical defect — Nanofat-seeded biological scaffold in healing larger surgical defects (>1.5cm) involving the lower limbs
  Arms: Nanofat-seeded biological scaffold on surgical defect

SUMMARY:
Large full-thickness skin defects, such as those resulting from trauma, large and giant congenital nevi, disfiguring scars, or tumor resection remain major clinical problems to patients and physicians. Skin flaps and grafts represent the current standard of care (SOC), but often present limitations associated with surgical morbidity and donor site availability. The investigators will enroll 64 patients who have their skin cancer surgically removed and require reconstructive procedure such as a skin flap/graft.

To objective of this study is to assess the efficacy and safety of a nanofat-seeded biological scaffold versus the SOC in healing larger surgical defects (>1.5cm) involving the lower limb that cannot be closed by direct suture and thus need a reconstructive procedure such as a skin flap/graft.

DETAILED DESCRIPTION:
Large full-thickness skin defects, such as those resulting from trauma, large and giant congenital nevi, disfiguring scars, or tumor resection remain major clinical problems to patients and physicians. Skin flaps and grafts represent the current standard of care (SOC), but often present limitations associated with surgical morbidity and donor site availability. To overcome these limitations, cultured epidermal autografts consisting of keratinocytes were developed to provide enough autologous skin. However, the routine use of these cultured epidermal autografts was hampered by its high risk of recurrent wound opening, long-term fragility, and increased rates of scar contractures.

Tissue-engineered dermal skin substitutes containing complex dermal layers have also been developed to produce large, near-natural skin substitutes. They promote healing and avoid scar contracture; however, the healing times are long as they lack the active cellular and paracrine components of healing, and they often need a second delayed surgical procedure, a split-thickness skin graft, to obtain complete epithelization.

The term "nanofat grafting" was first used by Tonnard et al. and constitutes a rich reservoir of regenerative precursor cells (including stromal vascular fraction cells, among which adipose-derived stem cells) with pro-angiogenic capabilities. The many proprieties of nanofat and the stromal vascular fraction in regenerative and aesthetic surgery are just being discovered. In particular, numerous in vitro and in vivo studies have demonstrated the ability of these cells to differentiate into various skin cell lineages. Moreover, they are recognized as a powerful source for tissue regeneration because of their capability to secrete paracrine factors, initiating tissue repair and accelerating wound closure by skin regeneration instead of fibrotic scar formation.

Few anecdotal reports have documented the efficacy of the stromal vascular fraction in acute as well as chronic wounds. However, no observation has explored the efficacy of nanofat in healing surgical defects. Of note, nanofat is substantially easier, faster, and remarkably less expensive to obtain when compared to the mechanically- or enzymatically-isolated stromal vascular fraction. At present, there is a noticeable lack of randomized-controlled evidence in the international literature. Thus, this would represent the most comprehensive and the first randomized, controlled experience documenting the use of nanofat for wound healing.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who need to undergo a surgical intervention resulting in complex lower limb surgical defects that cannot be closed primarily, and thus need a reconstructive phase
* Willing to undertake all study procedures, including nanofat harvesting from stomach site
* Willing to sign an informed consent form

Exclusion Criteria:

* Age less than 18 years of age
* Pregnant women
* Any contraindications to use of nanofat or collagen scaffold

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in healing response to treatment (>95% healed in surface by physician assessment) | 7 days post-surgery, 15 days post-surgery, 30 days post-surgery, 3 months post-surgery, 6 months post-surgery, 12 months post-surgery
  A blinded study physician will assess the healing surface area at each visit. A wound is considered "healed" when the wound has healed >95% in surface by the physician assessment. Wounds in the intervention group are expected to have faster healing compared to the standard of care group.

SECONDARY OUTCOMES:
Change in histogram planimetry for surgical site | 7 days' post-surgery, 15 days' post-surgery, 30 days' post-surgery, 3 months' post-surgery, 6 months' post-surgery, 12 months' post-surgery
  Histogram planimetry is a way to objectively assess wound area changes over time. It is based on the pixel count of a selected irregular area which is divided by the pixel count of 1cm^2 to find a result in terms of cm^2 or mm^2
Cosmetic outcomes of surgical site by blinded physician Vancouver Scar Scale assessment | 3 months' post-surgery, 6 months' post-surgery
  A physician blinded to the treatment group the subject is in will self-administer the Vancouver Scar Scale (VSS) which documents change in scar appearance over time. The VSS ranges from 0 (most desirable outcome) to 13 (least desirable outcome), thus, a lower score is considered to have a better outcome and a higher score is considered a worse outcome. The VSS consists of four sub-scales, with each sub-scale reporting a value. The "pigmentation sub-scale" ranges from 0 (normal pigmentation) to 2 (hyperpigmentation); the "vascularity sub-scale" ranges from 0 (normal appearance) to 3 (purple appearance); the "pliability sub-scale" ranges from 0 (normal pliability) to 5 (contracture); and the "height sub-scale" ranges from 0 (normal [flat]) to 3 (>5mm). Sub-scale scores are totaled to give an overall VSS assessment score.
Study subject completes the Patient Scar Assessment Scale | 3 months' post-surgery, 6 months' post-surgery
  Subjects will be asked to complete a Visual Analogue Scale (Patient Scar Assessment Scale, PSAS) for scar assessment to rate how they think their wound site appears cosmetically compared to normal skin, and any complaints about how painful the site is, and how itchy it feels. Each question ranges from 1 (no complaints with itch or pain/as normal skin) to 10 (worst imaginable itch or pain/very different from normal skin). The PSAS ranges from 6 (best outcome score) to 66 (worst outcome score), thus a lower score is considered to have a better outcome and a higher score is considered a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Chrysalyne D Schmults, MD, MSCE, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Mohs and Dermatologic Surgery Center, Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Klar AS, Zimoch J, Biedermann T. Skin Tissue Engineering: Application of Adipose-Derived Stem Cells. Biomed Res Int. 2017;2017:9747010. doi: 10.1155/2017/9747010. Epub 2017 Feb 27. PMID 28337463
- [Background] Tonnard P, Verpaele A, Peeters G, Hamdi M, Cornelissen M, Declercq H. Nanofat grafting: basic research and clinical applications. Plast Reconstr Surg. 2013 Oct;132(4):1017-1026. doi: 10.1097/PRS.0b013e31829fe1b0. PMID 23783059
- [Background] Cervelli V, Gentile P, De Angelis B, Calabrese C, Di Stefani A, Scioli MG, Curcio BC, Felici M, Orlandi A. Application of enhanced stromal vascular fraction and fat grafting mixed with PRP in post-traumatic lower extremity ulcers. Stem Cell Res. 2011 Mar;6(2):103-11. doi: 10.1016/j.scr.2010.11.003. Epub 2010 Nov 30. PMID 21195687
- [Background] You HJ, Han SK. Cell therapy for wound healing. J Korean Med Sci. 2014 Mar;29(3):311-9. doi: 10.3346/jkms.2014.29.3.311. Epub 2014 Feb 27. PMID 24616577
- [Background] Konstantinow A, Arnold A, Djabali K, Kempf W, Gutermuth J, Fischer T, Biedermann T. Therapy of ulcus cruris of venous and mixed venous arterial origin with autologous, adult, native progenitor cells from subcutaneous adipose tissue: a prospective clinical pilot study. J Eur Acad Dermatol Venereol. 2017 Dec;31(12):2104-2118. doi: 10.1111/jdv.14489. Epub 2017 Sep 4. PMID 28750144
- [Background] Brett E, Chung N, Leavitt WT, Momeni A, Longaker MT, Wan DC. A Review of Cell-Based Strategies for Soft Tissue Reconstruction. Tissue Eng Part B Rev. 2017 Aug;23(4):336-346. doi: 10.1089/ten.TEB.2016.0455. Epub 2017 Apr 27. PMID 28372485
- [Background] Klinger A, Kawata M, Villalobos M, Jones RB, Pike S, Wu N, Chang S, Zhang P, DiMuzio P, Vernengo J, Benvenuto P, Goldfarb RD, Hunter K, Liu Y, Carpenter JP, Tulenko TN. Living scaffolds: surgical repair using scaffolds seeded with human adipose-derived stem cells. Hernia. 2016 Feb;20(1):161-70. doi: 10.1007/s10029-015-1415-0. Epub 2015 Nov 6. PMID 26545361
- [Background] Uyulmaz S, Sanchez Macedo N, Rezaeian F, Giovanoli P, Lindenblatt N. Nanofat Grafting for Scar Treatment and Skin Quality Improvement. Aesthet Surg J. 2018 Mar 14;38(4):421-428. doi: 10.1093/asj/sjx183. PMID 29365061